CLINICAL TRIAL: NCT00819585
Title: A 24-week, Dose-ranging, Multicenter, Double-blind, Double-dummy, Active-controlled Core Study to Evaluate Canakinumab for Prophylaxis of Signs and Symptoms of Acute Flares in Chronic Gout Patients Initiating Allopurinol Therapy and a 24-week Open-label, Multicenter Extension Study to Assess Safety, Tolerability and Efficacy of Canakinumab in Patients With Gout Who Are Given Canakinumab at the Time of Gout Flare
Brief Title: A Study of the Efficacy of Canakinumab in Prevention of Acute Flares in Chronic Gout Patients Initiating Allopurinol Therapy (Core Study) and a Long-term Study of the Efficacy and Safety of Canakinumab in Patients With Gout (Extension Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CACZ885H2251; EudraCT : 2008-005876-28
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Gout
Keywords: Gout; Chronic gout; Gouty arthritis; Gout flares
MeSH Terms: conditions — Gout; Arthritis, Gouty | interventions — canakinumab; Colchicine; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (11):
- Core study: Canakinumab 25 mg (Experimental): Canakinumab 25 mg subcutaneously (sc) once at Day 1, placebo sc at Days 29, 57, and 85 plus daily placebo capsules for 16 weeks. Allopurinol treatment was initiated at the latest at baseline (Visit 2) according to the patient's renal function / estimated creatinine clearance at screening (Visit 1). Allopurinol was administered orally to all randomized patients once daily (100 mg-300 mg) for 24 weeks.
  Interventions: Drug: Canakinumab; Drug: Allopurinol; Drug: Placebo Matching Canakinumab; Drug: Placebo Matching Colchicine
- Core study: Canakinumab 50 mg (Experimental): Canakinumab 50 mg sc once at Day 1, placebo sc at Days 29, 57, and 85 plus daily placebo capsules for 16 weeks. Allopurinol treatment was initiated at the latest at baseline (Visit 2) according to the patient's renal function / estimated creatinine clearance at screening (Visit 1). Allopurinol was administered orally to all randomized patients once daily (100 mg-300 mg) for 24 weeks.
  Interventions: Drug: Canakinumab; Drug: Allopurinol; Drug: Placebo Matching Canakinumab; Drug: Placebo Matching Colchicine
- Core study: Canakinumab 100 mg (Experimental): Canakinumab 100 mg sc once at Day 1, placebo sc at Days 29, 57, and 85 plus daily placebo capsules for 16 weeks. Allopurinol treatment was initiated at the latest at baseline (Visit 2) according to the patient's renal function / estimated creatinine clearance at screening (Visit 1). Allopurinol was administered orally to all randomized patients once daily (100 mg-300 mg) for 24 weeks.
  Interventions: Drug: Canakinumab; Drug: Allopurinol; Drug: Placebo Matching Canakinumab; Drug: Placebo Matching Colchicine
- Core study: Canakinumab 200 mg (Experimental): Canakinumab 100 mg sc once at Day 1, placebo sc at Days 29, 57, and 85 plus daily placebo capsules for 16 weeks. Allopurinol treatment was initiated at the latest at baseline (Visit 2) according to the patient's renal function / estimated creatinine clearance at screening (Visit 1). Allopurinol was administered orally to all randomized patients once daily (100 mg-300 mg) for 24 weeks.
  Interventions: Drug: Canakinumab; Drug: Allopurinol; Drug: Placebo Matching Canakinumab; Drug: Placebo Matching Colchicine
- Core study: Canakinumab 300 mg (Experimental): Canakinumab 300 mg sc once at Day 1, placebo sc at Days 29, 57, and 85 plus daily placebo capsules for 16 weeks. Allopurinol treatment was initiated at the latest at baseline (Visit 2) according to the patient's renal function / estimated creatinine clearance at screening (Visit 1). Allopurinol was administered orally to all randomized patients once daily (100 mg-300 mg) for 24 weeks.
  Interventions: Drug: Canakinumab; Drug: Allopurinol; Drug: Placebo Matching Canakinumab; Drug: Placebo Matching Colchicine
- Core study: Canakinumab q4wk (Experimental): Canakinumab 50 mg sc at Days 1, and 29 followed by canakinumab 25 mg sc on Days 57, and 85 plus daily placebo capsules for 16 weeks, repeated every 4 week (q4wk). Allopurinol treatment was initiated at the latest at baseline (Visit 2) according to the patient's renal function / estimated creatinine clearance at screening (Visit 1). Allopurinol was administered orally to all randomized patients once daily (100 mg-300 mg) for 24 weeks.
  Interventions: Drug: Canakinumab; Drug: Allopurinol; Drug: Placebo Matching Colchicine
- Core study: Colchicine 0.5 mg (Active Comparator): Colchicine 0.5 mg capsule orally once daily throughout the whole treatment phase of 16 weeks plus placebo matching canakinumab s.c. at Days 1, 29, 57, and 85. Allopurinol treatment was initiated at the latest at baseline (Visit 2) according to the patient's renal function / estimated creatinine clearance at screening (Visit 1). Allopurinol was administered orally to all randomized patients once daily (100 mg-300 mg) for 24 weeks.
  Interventions: Drug: Colchicine; Drug: Allopurinol; Drug: Placebo Matching Canakinumab
- Extension study: Group A (Experimental): Participants who were randomized to canakinumab in the core study and were treated with canakinumab for at least 1 flare in the extension study.
  Interventions: Drug: Canakinumab
- Extension study: Group B (Experimental): Patients who were randomized to canakinumab in the core study but did not receive treatment with canakinumab in the extension study.
  Interventions: Drug: Canakinumab
- Extension study: Group C (Experimental): Patients who were randomized to colchicine in the core study and were treated with canakinumab for at least 1 flare in the extension study.
  Interventions: Drug: Canakinumab; Drug: Colchicine
- Extension study: Group D (Experimental): Patients who were randomized to colchicine in the core study but did not receive treatment with canakinumab in the extension study.
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Canakinumab — Canakinumab was supplied in glass vials as a lyophilized powder.
  Arms: Core study: Canakinumab 100 mg; Core study: Canakinumab 200 mg; Core study: Canakinumab 25 mg; Core study: Canakinumab 300 mg; Core study: Canakinumab 50 mg; Core study: Canakinumab q4wk; Extension study: Group A; Extension study: Group B; Extension study: Group C
Drug: Colchicine — 0.5 mg capsule orally once daily for 16 weeks.
  Arms: Core study: Colchicine 0.5 mg; Extension study: Group C; Extension study: Group D
Drug: Allopurinol — 100-300 mg orally once daily for 24 weeks.
  Arms: Core study: Canakinumab 100 mg; Core study: Canakinumab 200 mg; Core study: Canakinumab 25 mg; Core study: Canakinumab 300 mg; Core study: Canakinumab 50 mg; Core study: Canakinumab q4wk; Core study: Colchicine 0.5 mg
Drug: Placebo Matching Canakinumab — Subcutaneous injection.
  Arms: Core study: Canakinumab 100 mg; Core study: Canakinumab 200 mg; Core study: Canakinumab 25 mg; Core study: Canakinumab 300 mg; Core study: Canakinumab 50 mg; Core study: Colchicine 0.5 mg
Drug: Placebo Matching Colchicine — Capsule orally once daily for 16 weeks.
  Arms: Core study: Canakinumab 100 mg; Core study: Canakinumab 200 mg; Core study: Canakinumab 25 mg; Core study: Canakinumab 300 mg; Core study: Canakinumab 50 mg; Core study: Canakinumab q4wk

SUMMARY:
The 24-week, dose-ranging, multi-center, double-blind, double-dummy, active-controlled core study investigated the prophylactic effect of canakinumab on the signs and symptoms of acute flares in chronic gout patients initiating allopurinol therapy. The core study was followed by a 24-week open-label, multicenter extension study to assess the safety, tolerability, and efficacy of canakinumab in patients with gout who were given canakinumab at the time of gout flare.

ELIGIBILITY:
Core study

Inclusion Criteria:

* Signed written informed consent before any study procedure is performed.
* History of at least 2 gout flares in the year prior to Screening (Visit 1, based on patient history), thus, candidates for initiating uric acid lowering therapy.
* Confirmed diagnosis of gout meeting the American College of Rheumatology (ACR) 1977 preliminary criteria for the classification of arthritis of primary gout.
* Body Mass Index (BMI) ≤ 40 kg/m^2.
* Willingness to initiate allopurinol therapy as urate lowering agent for their gout therapy or having initiated allopurinol therapy within ≤ 1 month before Screening (Visit 1) or willing to re-initiate allopurinol therapy if this was stopped > 2 months before Screening (Visit 1) for reasons different to toxicity/ intolerance or lack of efficacy.

Exclusion Criteria:

* Acute gout flare within 2 weeks of Screening (Visit 1) and during the Screening period.
* History of allergy or contraindication to colchicine or allopurinol.
* History of intolerance to allopurinol or to oral colchicine in appropriate dose for prophylactic use.
* History of bone marrow suppression.
* Absolute or relative contraindication to both naproxen and oral prednisolone/ prednisone.

Extension study

Inclusion criteria:

* Patients who completed the core study. A patient is defined as completing the core study if he/she completed the study up to and including the last visit (Visit 9).
* Patients who have signed a written informed consent before any trial procedure is performed.

Exclusion Criteria:

* Patients for whom continuation in the extension study is not considered appropriate by the treating physician.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive pregnancy test (serum or urine).

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2008-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (89):
- United States (19):
  - Talbert Medical Group, Huntington Beach, California
  - San Diego Arthritis & Osteoporosis Medical clinic, San Diego, California
  - Health Awareness, Jupiter, Florida
  - East-West Medical Research institute, Honolulu, Hawaii
  - Pinnacle Medical Research, Overland Park, Kansas
  - Cotton O'Neil Clinical Research Institute, Topeka, Kansas
  - Dolby Research, LLC, Baton Rouge, Louisiana
  - The Family Doctors, Shreveport, Louisiana
  - Shores Rheumatology, Saint Clair Shores, Michigan
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - NM Clinical Research & Osteoporosis Ct., Albuquerque, New Mexico
  - Rochester clinical Research, Rochester, New York
  - Health Research of Oklahoma, PLLC, Oklahoma City, Oklahoma
  - Castlerock Clinical Research Consultants, LLC, Tulsa, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Columbia Clinical Research, Columbia, South Carolina
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - MultiSpecialty Clinical Research, Johnson City, Tennessee
  - iMED Internal medicine, PA, San Antonio, Texas
- Argentina (3):
  - Novartis Investigative site, Buenos Aires
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative site, Rosario
- Belgium (2):
  - Novartis Investigative Site, Gozée
  - Novartis Investigative site, Oostham
- Colombia (4):
  - Novartis Investigative Site, Bacaramanga
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Fundación Cardiovascular de Colombia, Florida Blanca
- Czechia (5):
  - Novartis Investigative site, Havířov
  - Novartis Investigative site, Ostrava
  - Novartis Investigative site, Pardubice
  - Novartis Investigative site, Uherské Hradiště
  - Novartis Investigative site, Zlín
- Germany (12):
  - Novartis Investigative Site, Bautzen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Georgensgmünd
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Messkirch
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Riedlhuette
  - Novartis Investigative Site, Schwabach
- Novartis Investigative site, Guatemala City, Guatemala
- Hungary (4):
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Zalaegerszeg
- Poland (2):
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Wroclaw
- Portugal (3):
  - Novartis Investigative site, Coimbra
  - Novartis Investigative site, Lisbon
  - Novartis Investigative site, Ponte de Lima
- Russia (6):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative site, Moscow
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative site, Singapore, Singapore
- Slovakia (7):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Piešťany
  - Novartis Investigative Site, Považská Bystrica
  - Novartis Investigative site, Trebišov
- South Africa (3):
  - Novartis Investigative site, Cape Town
  - Novartis Investigative site, Panorama
  - Novartis Investigative site, Port Elizabeth
- Spain (4):
  - Novartis Investigative Site, Barakaldo
  - Novartis Investigative site, Madrid
  - Novartis Investigative site, Mérida
  - Novartis Investigative site, Valencia
- Taiwan (3):
  - Novartis Investigative site, Kaohsiung City
  - Novartis Investigative site, Taichung
  - Novartis Investigative site, Taipei
- Turkey (Türkiye) (8):
  - Baskent University Medical Faculty, Adana
  - Baskent University Medical Faculty, Ankara
  - Adnan Menderes University Medical Faculty, Aydin
  - Cukurova University Medical Faculty, Balcali Adana
  - Pamukkale University medical Faculty, Denizli Kampus
  - Gaziantep University Medical Faculty, Gaziantep
  - Dokuz Eylul University Medical Faculty, Izmir
  - Celal Bayar University Medical Faculty, Manisa
- United Kingdom (2):
  - Gables Medicentre, Coventry
  - Flyde Coast Clinical Research Ltd, Lancashire

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 432 participants were enrolled in the study.
Groups:
- Core Study: Canakinumab 25 mg: Participants received canakinumab 25 mg subcutaneously (sc) on Day 1; canakinumab placebo sc on Days 29, 57, and 85; and colchicine placebo orally once daily for 16 weeks.
- Core Study: Canakinumab 50 mg: Participants received canakinumab 50 mg sc on Day 1; canakinumab placebo sc on Days 29, 57, and 85; and colchicine placebo orally once daily for 16 weeks.
- Core Study: Canakinumab 100 mg: Participants received canakinumab 100 mg sc on Day 1; canakinumab placebo sc on Days 29, 57, and 85; and colchicine placebo orally once daily for 16 weeks.
- Core Study: Canakinumab 200 mg: Participants received canakinumab 200 mg sc on Day 1; canakinumab placebo sc on Days 29, 57, and 85; and colchicine placebo orally once daily for 16 weeks.
- Core Study: Canakinumab 300 mg: Participants received canakinumab 300 mg sc on Day 1; canakinumab placebo sc on Days 29, 57, and 85; and colchicine placebo orally once daily for 16 weeks.
- Core Study: Canakinumab q4wk: Participants received canakinumab 50 mg sc on Days 1 and 29; canakinumab 25 mg sc on Days 57 and 85; and colchicine placebo orally once daily for 16 weeks.
- Core Study: Colchicine 0.5 mg: Participants received colchicine 0.5 mg orally once daily for 16 weeks and canakinumab placebo sc on Days 1, 29, 57, and 85.
Period: Core Study
Arm/Group | Core Study: Canakinumab 25 mg | Core Study: Canakinumab 50 mg | Core Study: Canakinumab 100 mg | Core Study: Canakinumab 200 mg | Core Study: Canakinumab 300 mg | Core Study: Canakinumab q4wk | Core Study: Colchicine 0.5 mg | Extension Study: Group A | Extension Study: Group B | Extension Study: Group C | Extension Study: Group D
Started | 55 (Participants who started the core study are included in the randomized and full analysis sets.) | 54 | 54 | 54 | 53 | 54 | 108 | 0 (There were no participants in this arm during the core study.) | 0 (There were no participants in this arm during the core study.) | 0 (There were no participants in this arm during the core study.) | 0 (There were no participants in this arm during the core study.)
Received Study Medication | 55 (Participants who received study medication are included in the safety population.) | 54 | 54 | 54 | 53 | 53 (One participant in this treatment arm was HIV+ve and did not receive any study medication.) | 108 | 0 | 0 | 0 | 0
Completed | 49 | 48 | 48 | 49 | 50 | 52 | 95 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 5 | 3 | 2 | 13 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 1 | 4 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Abnormal Laboratory Value(s) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory Therapeutic Effect | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Subject No Longer Requires Study Drug | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject Withdrew Consent | 0 | 3 | 2 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Administrative Problems | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Period: Extension Study
Arm/Group | Core Study: Canakinumab 25 mg | Core Study: Canakinumab 50 mg | Core Study: Canakinumab 100 mg | Core Study: Canakinumab 200 mg | Core Study: Canakinumab 300 mg | Core Study: Canakinumab q4wk | Core Study: Colchicine 0.5 mg | Extension Study: Group A | Extension Study: Group B | Extension Study: Group C | Extension Study: Group D
Started | 0 (There were no participants in this arm during the extension study.) | 0 (There were no participants in this arm during the extension study.) | 0 (There were no participants in this arm during the extension study.) | 0 (There were no participants in this arm during the extension study.) | 0 (There were no participants in this arm during the extension study.) | 0 (There were no participants in this arm during the extension study.) | 0 (There were no participants in this arm during the extension study.) | 75 | 181 | 25 | 60
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 75 | 173 | 24 | 58
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 1 | 2
Not completed — Abnormal Laboratory Value(s) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Subject Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics of the reporting groups are based on the safety set, which included all participants who received study medication. Of the 432 participants enrolled in the core study, 1 participant did not receive any study medication and was not included in the safety set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Core Study: Canakinumab 25 mg | Core Study: Canakinumab 50 mg | Core Study: Canakinumab 100 mg | Core Study: Canakinumab 200 mg | Core Study: Canakinumab 300 mg | Core Study: Canakinumab q4wk | Core Study: Colchicine 0.5 mg | Total
Number analyzed (Participants) | 55 | 54 | 54 | 54 | 53 | 53 | 108 | 431
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.7 (9.72) | 54.4 (12.18) | 51.3 (12.41) | 52.6 (10.78) | 52.4 (11.30) | 52.8 (10.38) | 52.4 (10.69) | 52.4 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 6 | 4 | 2 | 4 | 7 | 26
  Male | 55 | 51 | 48 | 50 | 51 | 49 | 101 | 405

OUTCOME MEASURES:

1. Secondary Outcome: Core Study: Mean Number of Gout Flares for the Repeat Dose Regimen of Canakinumab as Compared to the Single Doses of Canakinumab
Time Frame: up to 16 weeks after randomization
Population: The Full Analysis Set (FAS) consisted of all patients as randomized that had at least 1 post-baseline assessment of the primary efficacy variable. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization.
Measure: Least Squares Mean (Standard Error); unit: gout flares per patient
Groups:
- Canakinumab 25 mg: Canakinumab 25 mg subcutaneously (s.c.) once at Day 1, placebo s.c. at Days 29, 57, and 85 plus daily placebo capsules for 16 weeks. Allopurinol treatment was initiated at the latest at baseline (Visit 2) according to the patient's renal function / estimated creatinine clearance at screening (Visit 1). Allopurinol was administered orally to all randomized patients once daily (100 mg- 300 mg) for 24 weeks.
- Canakinumab 50 mg: Canakinumab 50 mg s.c. once at Day 1, placebo s.c. at Days 29, 57, and 85 plus daily placebo capsules for 16 weeks. Allopurinol treatment was initiated at the latest at baseline (Visit 2) according to the patient's renal function / estimated creatinine clearance at screening (Visit 1). Allopurinol was administered orally to all randomized patients once daily (100 mg- 300 mg) for 24 weeks.
- Canakinumab 100 mg: Canakinumab 100 mg s.c. once at Day 1, placebo s.c. at Days 29, 57, and 85 plus daily placebo capsules for 16 weeks. Allopurinol treatment was initiated at the latest at baseline (Visit 2) according to the patient's renal function / estimated creatinine clearance at screening (Visit 1). Allopurinol was administered orally to all randomized patients once daily (100 mg- 300 mg) for 24 weeks.
- Canakinumab 200 mg: Canakinumab 200 mg s.c. once at Day 1, placebo s.c. at Days 29, 57, and 85 plus daily placebo capsules for 16 weeks. Allopurinol treatment was initiated at the latest at baseline (Visit 2) according to the patient's renal function / estimated creatinine clearance at screening (Visit 1). Allopurinol was administered orally to all randomized patients once daily (100 mg- 300 mg) for 24 weeks.
- Canakinumab 300 mg: Canakinumab 300 mg s.c. once at Day 1, placebo s.c. at Days 29, 57, and 85 plus daily placebo capsules for 16 weeks. Allopurinol treatment was initiated at the latest at baseline (Visit 2) according to the patient's renal function / estimated creatinine clearance at screening (Visit 1). Allopurinol was administered orally to all randomized patients once daily (100 mg- 300 mg) for 24 weeks.
- Canakinumab q4wk: Canakinumab 50 mg s.c. at Days 1, and 29 followed by canakinumab 25 mg s.c. on Days 57, and 85 plus daily placebo capsules for 16 weeks, repeated every 4 week (q4wk). Allopurinol treatment was initiated at the latest at baseline (Visit 2) according to the patient's renal function / estimated creatinine clearance at screening (Visit 1). Allopurinol was administered orally to all randomized patients once daily (100 mg- 300 mg) for 24 weeks.
Arm/Group | Canakinumab 25 mg | Canakinumab 50 mg | Canakinumab 100 mg | Canakinumab 200 mg | Canakinumab 300 mg | Canakinumab q4wk
Number analyzed (Participants) | 55 | 54 | 54 | 54 | 53 | 54
gout flares per patient | 0.48 (0.204) | 0.43 (0.207) | 0.22 (0.209) | 0.38 (0.205) | 0.21 (0.209) | 0.68 (0.209)

2. Secondary Outcome: Core Study: Percentage of Participants With at Least 1 Gout Flare Within 16 Weeks After Randomization
Description: The percentage of participants experiencing at least 1 gout flare within 16 weeks after randomization. A gout flare was defined as an increase in participant-reported gout pain in the most affected joint during a gout attack.
Time Frame: Baseline of the core study to Week 16
Population: Full Analysis Set (FAS): All patients as randomized that had at least 1 post-baseline assessment of the primary efficacy variable. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned at randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Core Study: Canakinumab 25 mg | Core Study: Canakinumab 50 mg | Core Study: Canakinumab 100 mg | Core Study: Canakinumab 200 mg | Core Study: Canakinumab 300 mg | Core Study: Canakinumab q4wk | Core Study: Colchicine 0.5 mg
Number analyzed (Participants) | 55 | 54 | 54 | 54 | 53 | 54 | 108
Percentage of participants | 27.3 | 16.7 | 14.8 | 18.5 | 15.1 | 16.7 | 44.4

3. Secondary Outcome: Core Study: Percentage of Participants With Gout Flare at Different Time Points
Description: A gout flare was defined as an increase in participant-reported gout pain in the most affected joint during a gout attack.
Time Frame: Days 2, 4, 6, and Weeks 2, 4, 6, 10, and 16 of the core study
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Core Study: Canakinumab 25 mg | Core Study: Canakinumab 50 mg | Core Study: Canakinumab 100 mg | Core Study: Canakinumab 200 mg | Core Study: Canakinumab 300 mg | Core Study: Canakinumab q4wk | Core Study: Colchicine 0.5 mg
Number analyzed (Participants) | 55 | 54 | 54 | 54 | 53 | 54 | 108
Percentage of participants
  2 days post-dose | 5.5 [1.79 to 15.96] | 3.7 [0.94 to 14.01] | 3.7 [0.94 to 14.01] | 3.7 [0.94 to 14.01] | 0.0 [0.0 to 0.0] | 3.8 [0.96 to 14.26] | 5.6 [2.53 to 11.95]
  4 days post-dose | 10.9 [5.05 to 22.68] | 3.7 [0.94 to 14.01] | 3.7 [0.94 to 14.01] | 3.7 [0.94 to 14.01] | 5.7 [1.86 to 16.53] | 3.8 [0.96 to 14.26] | 10.2 [5.77 to 17.64]
  6 days post-dose | 12.7 [6.28 to 24.85] | 5.6 [1.83 to 16.24] | 3.7 [0.94 to 14.01] | 7.4 [2.85 to 18.54] | 5.7 [1.86 to 16.53] | 3.8 [0.96 to 23.56] | 11.1 [6.47 to 18.74]
  2 weeks post-dose | 14.5 [7.55 to 26.99] | 7.4 [2.85 to 18.54] | 7.4 [2.85 to 18.54] | 11.1 [5.15 to 23.07] | 7.5 [2.90 to 18.87] | 11.3 [5.25 to 23.48] | 16.7 [10.85 to 25.14]
  4 weeks post-dose | 14.5 [7.55 to 26.99] | 9.3 [3.96 to 20.83] | 7.4 [2.85 to 18.54] | 13.0 [6.40 to 25.28] | 11.4 [5.27 to 23.56] | 15.1 [7.85 to 27.92] | 25.1 [17.93 to 34.38]
  6 weeks post-dose | 16.5 [8.96 to 29.39] | 11.1 [5.15 to 23.07] | 9.3 [3.98 to 20.91] | 13.0 [6.40 to 25.28] | 11.4 [5.27 to 23.56] | 27.92 [7.85 to 27.92] | 32.6 [24.58 to 42.30]
  10 weeks post-dose | 22.5 [13.43 to 36.26] | 13.1 [6.46 to 25.52] | 11.2 [5.19 to 23.22] | 16.8 [9.11 to 29.79] | 11.4 [5.27 to 23.56] | 17.0 [9.22 to 30.09] | 37.5 [29.06 to 47.43]
  16 weeks post-dose | 28.7 [18.34 to 43.10] | 17.3 [9.37 to 30.66] | 15.1 [7.82 to 27.87] | 18.8 [10.59 to 32.19] | 15.3 [7.96 to 28.29] | 17.0 [9.22 to 30.09] | 45.8 [36.76 to 55.87]

4. Secondary Outcome: Core Study: Participant's Assessment of Gout Pain on a 0-100 mm Visual Analog Scale up to Day 7 of All Gout Flares
Description: Participants rated the intensity of pain in the most affected joint on a 0-100 mm visual analog scale, which ranged from no pain (left end, 0) to unbearable pain (right end, 100). Participants assessed pain intensity on the day of onset of the gout flare and in the morning of the 6 following days.
Time Frame: Baseline of the core study to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Core Study: Canakinumab 25 mg | Core Study: Canakinumab 50 mg | Core Study: Canakinumab 100 mg | Core Study: Canakinumab 200 mg | Core Study: Canakinumab 300 mg | Core Study: Canakinumab q4wk | Core Study: Colchicine 0.5 mg
Number analyzed (Participants) | 55 | 54 | 54 | 54 | 53 | 54 | 108
Units on a scale
  Day 1 (n=15, 9, 8, 9, 8, 9, 48) | 41.1 (31.01) | 44.6 (15.82) | 56.3 (26.72) | 53.0 (27.99) | 52.2 (19.40) | 66.1 (15.07) | 53.1 (24.18)
  Day 2 (n=12, 7, 6, 5, 5, 7, 44) | 44.8 (30.06) | 40.1 (26.73) | 46.2 (35.11) | 19.8 (32.05) | 43.1 (17.62) | 59.3 (23.53) | 42.8 (24.37)
  Day 3 (n=10, 4, 4, 4, 4, 5, 38) | 31.5 (20.82) | 49.5 (18.48) | 49.5 (25.29) | 56.7 (40.91) | 26.3 (14.64) | 58.0 (27.59) | 38.1 (23.37)
  Day 4 (n=7, 3, 2, 3, 3, 6, 31) | 31.8 (16.77) | 46.3 (10.60) | 16.5 (23.33) | 63.5 (33.0) | 11.0 (11.0) | 49.4 (27.73) | 30.5 (26.68)
  Day 5 (n=7, 2, 1, 3, 2, 4, 22) | 19.3 (14.79) | 48.0 (5.66) | 0.0 (0.0) | 54.8 (43.38) | 13.0 (0.0) | 41.4 (33.63) | 31.8 (29.91)
  Day 6 (n=6, 1, 1, 2, 1, 3, 18) | 19.6 (14.14) | 44.0 (0.0) | 0.0 (0.0) | 57.5 (60.10) | 12.0 (0.0) | 43.5 (24.38) | 33.7 (26.66)
  Day 7 (n=6, 0, 1, 2, 1, 2, 16) | 20.9 (16.91) | NA (NA) — No data is available | 0.0 (0.0) | 35.0 (49.50) | 0.0 (0.0) | 52.0 (11.31) | 33.0 (22.16)

5. Secondary Outcome: Core Study: Participant's Assessment of Gout Pain on a 5-point Likert Scale up to Day 7 of All Gout Flares
Description: Participants assessed the intensity of pain in the most affected joint on a 5-point Likert scale, which ranged from 1 to 5 (1=None, 2=Mild, 3=Moderate, 4=Severe, 5=Extreme). Participants assessed pain intensity on the day of onset of the gout flare and in the morning of the 6 following days.
Time Frame: Baseline of the core study to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Core Study: Canakinumab 25 mg | Core Study: Canakinumab 50 mg | Core Study: Canakinumab 100 mg | Core Study: Canakinumab 200 mg | Core Study: Canakinumab 300 mg | Core Study: Canakinumab q4wk | Core Study: Colchicine 0.5 mg
Number analyzed (Participants) | 55 | 54 | 54 | 54 | 53 | 54 | 108
Units on a scale
  Day 1 (n=15, 8, 8, 9, 8, 9, 48) | 2.8 (0.88) | 3.1 (0.65) | 3.5 (1.20) | 3.2 (0.92) | 3.1 (0.35) | 3.8 (0.60) | 3.2 (0.77)
  Day 2 (n=12, 6, 6, 5, 5, 7, 44) | 2.9 (0.92) | 2.6 (1.02) | 3.3 (1.51) | 2.2 (1.10) | 2.9 (0.74) | 3.5 (1.05) | 3.0 (0.86)
  Day 3 (n=10, 4, 4, 4, 4, 6, 38) | 2.4 (0.73) | 3.1 (0.63) | 2.3 (0.96) | 3.0 (1.15) | 2.3 (0.50) | 3.4 (1.07) | 2.7 (0.76)
  Day 4 (n=7, 3, 2, 3, 3, 7, 31) | 2.6 (0.57) | 2.7 (0.58) | 1.5 (0.71) | 3.0 (1.00) | 1.7 (0.58) | 3.2 (1.08) | 2.4 (0.90)
  Day 5 (n=7, 2, 1, 3, 2, 4, 22) | 2.2 (0.69) | 2.5 (0.71) | 1.0 (0) | 3.2 (1.76) | 1.5 (0.71) | 2.7 (1.28) | 2.6 (0.95)
  Day 6 (n=6, 1, 1, 2, 2, 3, 18) | 2.4 (0.49) | 3.0 (0.0) | 1.0 (0.0) | 3.5 (2.12) | 1.5 (0.71) | 2.9 (0.84) | 2.5 (1.05)
  Day 7 (n=6, 0, 1, 2, 1, 2, 16) | 2.4 (0.49) | NA (NA) — No participants analyzed. | 1.0 (0.0) | 2.5 (2.12) | 1.0 (0.0) | 3.3 (0.47) | 2.4 (0.81)

6. Primary Outcome: Core Study: Mean Number of Gout Flares Per Participant
Description: as for outcome 3
Time Frame: Baseline of the core study to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Gout flares
Arm/Group | Core Study: Canakinumab 25 mg | Core Study: Canakinumab 50 mg | Core Study: Canakinumab 100 mg | Core Study: Canakinumab 200 mg | Core Study: Canakinumab 300 mg | Core Study: Canakinumab q4wk | Core Study: Colchicine 0.5 mg
Number analyzed (Participants) | 55 | 54 | 54 | 54 | 53 | 54 | 108
Gout flares | 0.5 (1.03) | 0.4 (1.82) | 0.2 (0.53) | 0.4 (1.35) | 0.2 (0.53) | 0.7 (2.24) | 0.7 (1.00)

7. Secondary Outcome: Core Study: Physician's Global Assessment of Response to Therapy on a 5-point Likert Scale
Description: The study physician made a global assessment of the participant's response to treatment on a 5-point Likert scale (Very good, Good, Fair, Poor, Very poor) at Days 15, 29, 57, 85, 113, and 141. The category 'Not assessed' includes missing data and 'not done'. The number of participants in each of the 5 categories of the Likert scale are reported.
Time Frame: Days 15, 29, 57, 85, 113, and 141 of the core study
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Core Study: Canakinumab 25 mg | Core Study: Canakinumab 50 mg | Core Study: Canakinumab 100 mg | Core Study: Canakinumab 200 mg | Core Study: Canakinumab 300 mg | Core Study: Canakinumab q4wk | Core Study: Colchicine 0.5 mg
Number analyzed (Participants) | 55 | 54 | 54 | 54 | 53 | 54 | 108
Participants
  Day 15: Very good | 19 | 23 | 24 | 23 | 27 | 25 | 40
  Day 15 - Good | 28 | 24 | 23 | 26 | 21 | 20 | 42
  Day 15 - Fair | 5 | 4 | 3 | 4 | 0 | 3 | 16
  Day 15 - Poor | 0 | 0 | 2 | 0 | 3 | 4 | 6
  Day 15 - Very poor | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Day 15 - Not assessed | 3 | 1 | 1 | 1 | 1 | 2 | 2
  Day 29: Very good | 26 | 24 | 25 | 24 | 27 | 27 | 39
  Day 29- Good | 23 | 22 | 22 | 26 | 23 | 22 | 42
  Day 29 - Fair | 2 | 4 | 5 | 3 | 2 | 2 | 19
  Day 29 - Poor | 0 | 0 | 1 | 0 | 0 | 2 | 2
  Day 29 - Very poor | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Day 29 - Not assessed | 0 | 3 | 0 | 0 | 0 | 1 | 3
  Day 57: Very good | 25 | 27 | 28 | 27 | 30 | 28 | 46
  Day 57- Good | 21 | 20 | 16 | 21 | 18 | 20 | 43
  Day 57 - Fair | 5 | 3 | 6 | 4 | 4 | 3 | 9
  Day 57 - Poor | 0 | 0 | 2 | 0 | 0 | 2 | 3
  Day 57 - Very poor | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Day 57 - Not assessed | 0 | 2 | 1 | 0 | 0 | 1 | 4
  Day 85: Very good | 27 | 31 | 32 | 32 | 31 | 29 | 43
  Day 85 - Good | 20 | 17 | 15 | 16 | 17 | 17 | 41
  Day 85 - Fair | 3 | 2 | 5 | 4 | 2 | 3 | 12
  Day 85 - - Poor | 0 | 0 | 1 | 0 | 1 | 2 | 2
  Day 85 - Very poor | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Day 85 - Not assessed | 1 | 2 | 0 | 0 | 1 | 1 | 5
  Day 113 : Very good | 24 | 29 | 30 | 26 | 29 | 32 | 50
  Day 113 - Good | 18 | 18 | 18 | 20 | 20 | 15 | 36
  Day 113 - Fair | 5 | 3 | 2 | 3 | 1 | 3 | 7
  Day 113 - Poor | 2 | 0 | 1 | 1 | 1 | 2 | 2
  Day 113 - Very poor | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Day 113 - Not Assessed | 0 | 2 | 0 | 0 | 0 | 2 | 8
  Day 141 : Very good | 26 | 25 | 24 | 31 | 32 | 32 | 41
  Day 141 - Good | 16 | 20 | 19 | 12 | 14 | 14 | 36
  Day 141 - Fair | 6 | 2 | 3 | 6 | 2 | 3 | 16
  Day 141 - Poor | 1 | 1 | 3 | 0 | 0 | 2 | 2
  Day 141 - Very poor | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Day 141 - Not Assessed | 0 | 3 | 1 | 0 | 1 | 1 | 5

8. Secondary Outcome: Extension Study: Participant's Assessment of Gout Pain on a 100 mm Visual Analog Scale During the First Flare
Description: Participant's rated the intensity of pain in the most affected joint during the first flare on a 0-100 mm visual analog scale, which ranged from no pain (left end, 0) to unbearable pain (right end, 100). Assessments were made pre-dose and 24 hours, 3 days, 4 days, and an average of 5-7 days post-dose
Time Frame: Baseline of the extension study until 7 days after the onset of the first gout flare (up to 24 weeks)
Population: Efficacy set: All Group A and C participants who received at least 1 dose of canakinumab during the extension study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Extension Study: Group A | Extension Study: Group C
Number analyzed (Participants) | 65 | 19
Units on a scale
  Pre-dose (n=65, 19) | 61.3 (27.13) | 71.8 (20.86)
  24 hours (n=65, 18) | 23.8 (23.32) | 29.0 (22.85)
  3 days (n=54, 15) | 12.4 (16.82) | 6.8 (9.03)
  4 days (n=54, 15) | 8.8 (14.32) | 2.7 (5.06)
  5-7 days (n=52, 13) | 8.1 (15.86) | 2.1 (4.70)

9. Secondary Outcome: Extension Study: Participant's Global Assessment of Response to Treatment on a 5-point Likert Scale
Description: Study participants made a global assessment of their response to treatment on a 5-point Likert scale (Excellent, Good, Acceptable, Slight, Poor) at the control visit 7±2 days following each of their first 3 flares. The number of participants in each of the 5 categories of the Likert scale are reported.
Time Frame: Baseline of the extension study until the end of the study (up to 24 weeks)
Population: Efficacy set: All Group A and C participants who received at least 1 dose of canakinumab during the extension study.
Measure: Number; unit: Participants
Arm/Group | Extension Study: Group A | Extension Study: Group C
Number analyzed (Participants) | 63 | 21
Participants
  Gout Flare 1: Excellent (63, 21) | 40 | 7
  Gout Flare 1: Good (63, 21) | 17 | 14
  Gout Flare 1: Acceptable (63, 21) | 5 | 0
  Gout Flare 1: Slight (63, 21) | 1 | 0
  Gout Flare 1: Poor (63, 21) | 0 | 0
  Gout Flare 2: Excellent (11, 5) | 4 | 4
  Gout Flare 2: Good (11, 5) | 6 | 1
  Gout Flare 2: Acceptable (11, 5) | 1 | 0
  Gout Flare 2: Slight (11, 5) | 0 | 0
  Gout Flare 2: Poor (11, 5) | 0 | 0
  Gout Flare 3: Excellent (3, 1) | 2 | 0
  Gout Flare 3: Good (3, 1) | 1 | 1
  Gout Flare 3: Acceptable (3, 1) | 0 | 0
  Gout Flare 3: Slight (3, 1) | 0 | 0
  Gout Flare 3: Poor (3, 1) | 0 | 0

10. Secondary Outcome: Extension Study: Physician's Global Assessment of Response to Treatment on a 5-point Likert Scale
Description: The study physician made a global assessment of the participant's response to treatment on a 5-point Likert scale (Very good, Good, Fair, Poor, Very poor) at the control visit 7±2 days following each of the first 3 flares. The category 'Not assessed' includes missing data and 'not done'. The number of participants in each of the 5 categories of the Likert scale are reported.
Time Frame: Baseline of the extension study until the end of the study (up to 24 weeks)
Population: Efficacy set: All Group A and C participants who received at least 1 dose of canakinumab during the extension study.
Measure: Number; unit: Participants
Arm/Group | Extension Study: Group A | Extension Study: Group C
Number analyzed (Participants) | 69 | 23
Participants
  Gout Flare 1: Very Good (69, 23) | 37 | 13
  Gout Flare 1: Good (69, 23) | 28 | 10
  Gout Flare 1: Fair (69, 23) | 2 | 0
  Gout Flare 1: Poor (69, 23) | 2 | 0
  Gout Flare 1: Very Poor (69, 23) | 0 | 0
  Gout Flare 2: Very Good (12, 5) | 5 | 3
  Gout Flare 2: Good (12, 5) | 7 | 2
  Gout Flare 2: Fair (12, 5) | 0 | 0
  Gout Flare 2: Poor (12, 5) | 0 | 0
  Gout Flare 2: Very Poor (12, 5) | 0 | 0
  Gout Flare 3: Very Good (3, 1) | 1 | 0
  Gout Flare 3: Good (3, 1) | 2 | 1
  Gout Flare 3: Fair (3, 1) | 0 | 0
  Gout Flare 3: Poor (3, 1) | 0 | 0
  Gout Flare 3: Very Poor (3, 1) | 0 | 0

11. Secondary Outcome: Extension Study: Physician's Assessment of Tenderness, Swelling, and Erythema in the Most Affected Joint During the First Flare
Description: Tenderness was rated on a 0-3 point scale: 0="no pain", 1=patient states that "there is pain", 2=patient states "there is pain and winces", and 3=patient states "there is pain, winces and withdraws" on palpation or passive movement of the most affected joint. Swelling was rated on a 0-3 point scale: 0="no swelling", 1="palpable", 2="visible", and 3=bulging beyond the joint margins". Erythema was rated as present, absent, or not assessable. Assessments were performed at the flare and control visits.
Time Frame: Baseline of the extension study until the end of the study (up to 24 weeks)
Population: Efficacy set: All Group A and C participants who received at least 1 dose of canakinumab during the extension study.
Measure: Number; unit: Participants
Arm/Group | Extension Study: Group A | Extension Study: Group C
Number analyzed (Participants) | 69 | 24
Participants
  Tenderness Flare Visit: No pain | 2 | 0
  Tenderness Flare Visit: Pain | 27 | 2
  Tenderness Flare Visit: Pain and winces | 23 | 10
  Tenderness Flare Visit: Pain, winces and withdraws | 17 | 12
  Tenderness Control Visit: No pain | 60 | 21
  Tenderness Control Visit: Pain | 8 | 3
  Tenderness Control Visit: Pain and winces | 1 | 0
  Tenderness Control Visit: Pain, winces and withdra | 0 | 0
  Joint Swelling Flare Visit: No swelling | 5 | 0
  Joint Swelling Flare Visit: Palpable | 20 | 2
  Joint Swelling Flare Visit: Visible | 31 | 17
  Joint Swelling Flare Visit: Bulging beyond joint | 13 | 5
  Joint Swelling Control Visit: No swelling | 61 | 22
  Joint Swelling Control Visit: Palpable | 6 | 2
  Joint Swelling Control Visit: Visible | 2 | 0
  Joint Swelling Control Visit: Bulging beyond joint | 0 | 0
  Erythema Flare Visit: Absent | 21 | 4
  Erythema Flare Visit: Present | 44 | 20
  Erythema Flare Visit: Not assessed | 0 | 0
  Erythema Control Visit: Absent | 66 | 24
  Erythema Control Visit: Present | 3 | 0
  Erythema Control Visit: Not assessed | 0 | 0

12. Secondary Outcome: Extension Study: Amount of Rescue Medication Taken
Description: The amount of naproxen and prednisolone taken after receiving treatment for each of the first 3 flares was recorded.
Time Frame: Baseline of the extension study until the end of the study (up to 24 weeks)
Population: Efficacy set: All Group A and C participants who received at least 1 dose of canakinumab during the extension study.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Extension Study: Group A | Extension Study: Group C
Number analyzed (Participants) | 68 | 24
mg
  Gout Flare 1: Naproxen (n=68, 24) | 1086.8 (1592.72) | 954.6 (1130.19)
  Gout Flare 1: Prednisolone (68, 24) | 4.6 (20.84) | 4.2 (20.41)
  Gout Flare 2: Naproxen (n=12, 5) | 650.0 (642.79) | 200.0 (447.21)
  Gout Flare 2: Prednisolone (12, 5) | 1.3 (3.11) | 0.0 (0.00)
  Gout Flare 3: Naproxen (n=4, 1) | 250.0 (500.00) | 0.0 (0.00)
  Gout Flare 3: Prednisolone (4, 1) | 0.0 (0.00) | 0.0 (0.00)

ADVERSE EVENTS:
Groups:
- Core Study: ACZ 25 mg: Core study: ACZ 25 mg
- Core Study: ACZ 50 mg: Core study: ACZ 50 mg
- Core Study: ACZ 100 mg: Core study: ACZ 100 mg
- Core Study: ACZ 200 mg: Core study: ACZ 200 mg
- Core Study: ACZ 300 mg: Core study: ACZ 300 mg
- Core Study: ACZ Q4wk mg: Core study: ACZ Q4wk mg
- Core Study: Colch 0.5 mg: Core study: Colch 0.5 mg
- Extension Study: Group A: Extension study: Group A
- Extension Study: Group B: Extension study: Group B
- Extension Study: Group C: Extension study: Group C
- Extension Study: Group D: Extension study: Group D
Arm/Group | Core Study: ACZ 25 mg | Core Study: ACZ 50 mg | Core Study: ACZ 100 mg | Core Study: ACZ 200 mg | Core Study: ACZ 300 mg | Core Study: ACZ Q4wk mg | Core Study: Colch 0.5 mg | Extension Study: Group A | Extension Study: Group B | Extension Study: Group C | Extension Study: Group D
Serious Adverse Events (participants affected / at risk) | 2/55 | 2/54 | 3/54 | 3/54 | 3/53 | 1/53 | 6/108 | 4/75 | 6/181 | 0/25 | 1/60
Other Adverse Events (participants affected / at risk) | 21/55 | 15/54 | 14/54 | 14/54 | 15/53 | 14/53 | 21/108 | 21/75 | 19/181 | 6/25 | 4/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Study: ACZ 25 mg (N=55) | Core Study: ACZ 50 mg (N=54) | Core Study: ACZ 100 mg (N=54) | Core Study: ACZ 200 mg (N=54) | Core Study: ACZ 300 mg (N=53) | Core Study: ACZ Q4wk mg (N=53) | Core Study: Colch 0.5 mg (N=108) | Extension Study: Group A (N=75) | Extension Study: Group B (N=181) | Extension Study: Group C (N=25) | Extension Study: Group D (N=60)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial fibrosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stupor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Study: ACZ 25 mg (N=55) | Core Study: ACZ 50 mg (N=54) | Core Study: ACZ 100 mg (N=54) | Core Study: ACZ 200 mg (N=54) | Core Study: ACZ 300 mg (N=53) | Core Study: ACZ Q4wk mg (N=53) | Core Study: Colch 0.5 mg (N=108) | Extension Study: Group A (N=75) | Extension Study: Group B (N=181) | Extension Study: Group C (N=25) | Extension Study: Group D (N=60)
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2 | 3 | 1 | 0 | 2 | 2 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2 | 2 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2 | 3 | 1 | 3 | 4 | 5 | 4 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 4 | 2 | 3 | 2 | 3 | 4 | 6 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 3 | 0 | 0 | 4 | 1 | 2 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 1 | 2 | 6 | 3 | 6 | 3 | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 4 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 6 | 2 | 2 | 5 | 4 | 2 | 1 | 6 | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.